CLINICAL TRIAL: NCT05427188
Title: Effect of Acute Psychosocial Stress on Esophageal Sensitivity in Healthy Volunteers
Brief Title: Effect of MIST on Esophageal Sensitivity in HV
Acronym: MIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: S65302-HV
Record Dates: First submitted 2021-10-20; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIST-paradigm (Experimental): HV assigned in the MIST paradigm will receive psychosocial stress
  Interventions: Behavioral: Stress paradigm
- Sham-paradigm (Sham Comparator): HV assigned in the MIST paradigm will receive no psychosocial stress
  Interventions: Behavioral: Sham paradigm

INTERVENTIONS:
Behavioral: Stress paradigm — HV will receive mental arithmetic challenges, together with social evaluative threat components from the program and/or the investigator
  Arms: MIST-paradigm
Behavioral: Sham paradigm — HV will receive mental arithmetic challenges where threat components from the program and/or the investigator are absent
  Arms: Sham-paradigm

SUMMARY:
Effect of acute psychosocial stress on esophageal sensitivity in healthy volunteers.

DETAILED DESCRIPTION:
Gastro-esophageal reflux disease (GERD), defined as the presence of symptoms or lesions that can be attributed to the reflux of gastric contents into the esophagus, is an increasingly prevalent condition in Western societies. The most typical symptoms are heartburn and regurgitation, however GERD can also manifest itself through a variety of other esophageal and extra-esophageal symptoms (e.g. chronic cough).

GERD patients can be divided into different categories based on upper endoscopy and pH or impedance-pH (MII-pH) monitoring. In the absence of lesions (esophagitis) during upper endoscopy, a pH or MII-pH monitoring will be performed. A first subcategory are patients with true GERD, characterized by an abnormal acid exposure and a positive or negative symptom association. The second and third category are patients with reflux hypersensitivity (RHS) and functional heartburn (FH)characterized by normal acid exposure on the MII-pH monitoring and a positive and negative symptom reflux association, respectively.

The basis for symptom generation/perception in GERD patients is not yet completely understood, but different mechanisms have been proposed including esophageal hypersensitivity, in which psychosocial stress is considered as a potential factor. This was shown in a study where 64% of the participants with heartburn reported that psychological factors, such as life stress, aggravate their symptoms. Furthermore, Fass et al. observed that auditory stress exacerbated symptom perception during esophageal acid perfusion (6). Moreover, our group investigated the effect of intravenous corticotrophin releasing hormone (CRH) on esophageal in healthy volunteers and showed that CRH is able to increase esophageal sensitivity to mechanical distention. Nevertheless, these previously performed studies in patients have some limitations: no measurable increase in cortisol (hypothalamo-pituitary-adrenal (HPA)-axis was not affected in these studies) and patients with RHS and FH - in whom the effect of stress is hypothesized to be the most relevant - were not included.

To induce moderate psychologic stress in the current study, the Montreal Imaging Stress Task (MIST) will be used. During this protocol, participants receive mental arithmetic challenges, together with social evaluative threat components from the program and/or the investigator (sham condition: threat components from the program and/or the investigator are absent). This MIST protocol can be used when investigating the effects of perceiving and processing psychosocial stress in the human brain in functional imaging studies.

Therefore, we want to investigate the relation between sensitivity to different stimuli (esophageal sensitivity) and psychosocial stress in healthy volunteers and patients (True GERD, RHS and FH).

ELIGIBILITY:
Inclusion Criteria:

Aged between 18 to 65 years. All participants will receive and sign a copy of the informed consent before initiation of the study.

Exclusion Criteria:

* A history of any upper gastrointestinal (GI) symptoms, complaints or diseases;
* Prior history of esophageal or gastric surgery or endoscopic anti-reflux procedure;
* Psychiatric disorders;
* Concomitant use of other medication or treatments except for oral contraceptives;
* Use of medication altering GI motility;
* Pregnant or nursing women;
* History of drugs or alcohol abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Esophageal mechanical sensitivity | Will be assessed at time point 180 minutes
  Change in balloon distention
Esophageal chemical sensitivity | We be assessed at time point 180 minutes
  Change in time for reaching pain threshold

SECONDARY OUTCOMES:
Cortisol levels | every 15 minutes a saliva sample during 4.5 hours: at time points (in minutes) 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240, 255, 27
  Change in cortisol levels

CONTACTS AND LOCATIONS:
Locations (1):
- TARGID, Leuven, Vlaams-Brabant, Belgium